CLINICAL TRIAL: NCT06071858
Title: Cluster Randomized Trial of Enhanced Coordinated Specialty Care (CSC 2.0) for Early Psychosis
Brief Title: Enhanced Coordinated Specialty Care for Early Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Boston Medical Center (Other); Cambridge Health Alliance (Other); University of Massachusetts, Worcester (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dost Ongur, Director, LEAP Center, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023P002612; 2P50MH115846-05 (NIH)
Record Dates: First submitted 2023-09-26; First posted 2023-10-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Psychosis; Schizophrenia; Schizoaffective Disorder; Psychosis Nos/Other; Bipolar Disorder
Keywords: first episode psychosis; early psychosis
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Bipolar Disorder | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coordinated Specialty Care (CSC; standard of care) (No Intervention): Care as usual; no intervention.
- Enhanced Coordinated Speciality Care (CSC 2.0) (Experimental): CSC 2.0 arm will be offered 1:1 peer support, digital outreach, care coordination, multi-family group therapy, and cognitive remediation (if applicable).
  Interventions: Behavioral: Care Coordination; Behavioral: Individual Peer Support; Behavioral: Digital Outreach; Behavioral: Cognitive Remediation; Behavioral: Multi-Family Group Therapy

INTERVENTIONS:
Behavioral: Care Coordination — * The study staff clinician will review all medical issues for each patient and reach out to primary care providers (PCP), dieticians, and other medical providers as needed.
  * The study staff clinician will serve as point person for communication with emergency departments and inpatient providers if the patient requires those levels of care.
  * The clinician will communicate with outside providers to provide background and ensure health decision making by those providers, visit and support patients as appropriate, access outside records and share with rest of the care team, and most critically ensure that a proper discharge plan has been made for the patient including care appointments, access to prescriptions and any new referrals made during hospitalization.
  Arms: Enhanced Coordinated Speciality Care (CSC 2.0)
Behavioral: Individual Peer Support — • Patients will be offered weekly 1:1 sessions with a Peer Provider as part of routine care in a mixture of in-person and virtual formats as appropriate to support patients around treatment decisions, and recovery.
  Arms: Enhanced Coordinated Speciality Care (CSC 2.0)
Behavioral: Digital Outreach — • mindLAMP smartphone application for various kinds of outreach including but not limited to medication and/or appointment reminders, resources, and activities such as breathing and meditation exercises.
  Arms: Enhanced Coordinated Speciality Care (CSC 2.0)
Behavioral: Cognitive Remediation — * For participants identified as needing and/or wanting support around cognition.
  * The cognitive remediation program is available online or in-app and offers memory, attention, processing speed, executive functioning, and social cognition training activities.
  Arms: Enhanced Coordinated Speciality Care (CSC 2.0)
Behavioral: Multi-Family Group Therapy — * Families whose loved ones are in CSC clinic will be offered weekly group sessions with a study staff clinician.
  * Each group may include 5-8 families and include a mixture of in-person and virtual formats.
  * These groups will be open-ended, including psychoeducation, and practical problem-solving discussions around care and other topics.
  Arms: Enhanced Coordinated Speciality Care (CSC 2.0)

SUMMARY:
The goal of this clinical trial is to compare engagement in treatment in coordinated specialty care (CSC) to five extra care elements (CSC 2.0) in first-episode psychosis. The main question it aims to answer is:

• Does the addition of certain elements of care increase the number of visits in treatment for first-episode psychosis?

Participants will either:

* Receive care as usual (CSC) or
* Receive care as usual (CSC) plus five additional care elements (CSC 2.0):

  1. Individual peer support
  2. Digital outreach
  3. Care coordination
  4. Multi-family group therapy
  5. Cognitive remediation

Researchers will compare the standard of care (CSC) to CSC 2.0 to see if participants receiving CSC 2.0 have more visits to their clinic in their first year.

ELIGIBILITY:
Inclusion Criteria:

* People undergoing an intake evaluation to CSC for first-episode psychosis in one of the following outpatient clinics:
* McLean Hospital OnTrack (OnTrack Clinic)
* Massachusetts General Hospital (FEPP Clinic)
* Boston Medical Center (WRAP Clinic)
* Cambridge Health Alliance (RISE Clinic)
* UMass Memorial Health Care (STEP Clinic)
* ServiceNet (PREP West)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Months Engaged in Care | 12 months following clinic intake
  Number of months each participant had ≥4 visits in a 12-month period

SECONDARY OUTCOMES:
Clinic Visit Number | 12 months following clinic intake
  Total number of clinic visits in a 12-month period
Clinic Visit Type | 12 months following clinic intake
  Numbers of different types of visits (eer provider, psychotherapy, psychopharmacology, group therapy, etc.) in a 12-month period
Duration of Treatment | Up to 12 months - measured as time between clinic intake and detachment
  Duration of time in treatment
Proportion in Arm Still in Clinic | 12 months following clinic intake
  Proportion of patients in each arm who are still in CSC at the end of the 12-month follow-up period

OTHER OUTCOMES:
Exploratory Analysis of symptom and functioning measures in EPINET Core Assessment Battery (CAB) | 12 months following clinic intake
  Exploratory analysis of variables collected by EPINET CAB by arm
Proportion of Early Detachment | 1 month
  Proportion of patients in each arm who detach from clinic prior to the end of their first month in care
Months Engaged in Care - extension of primary outcome | 24 months
  Number of months each participant had ≥4 visits in a 24-month period

CONTACTS AND LOCATIONS:
Overall Officials: Dost Ongur, MD, PhD, Principal Investigator — Mclean Hospital
Locations (5):
- United States (5):
  - McLean Hospital OnTrack Clinic, Belmont, Massachusetts
  - Massachusetts General Hospital FEPP Clinic, Boston, Massachusetts
  - Boston Medical Center WRAP, Boston, Massachusetts
  - Cambridge Health Alliance RISE Clinic, Cambridge, Massachusetts
  - UMass Memorial Community Healthlink STEP Clinic, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No